CLINICAL TRIAL: NCT03797235
Title: The Impact of Nerve Cross Section Area on Sensory Block Onset. A Prospective, Monocentric Crossover Study on Volunteers
Brief Title: The Impact of Nerve Cross Section Area on Sensory Block Onset
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Aguirre (Other)
Responsible Party: Sponsor-Investigator, Jose Aguirre, PD Dr. med., Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BASEC 2018-00939
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Regional Anesthesia
Keywords: Ultrasound-guided regional anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dominant Arm (Experimental): Two ultrasound guided nerve blocks (block of the ulnar and median nerve) on the dominant forearm
  Interventions: Procedure: Dominant Arm
- Non-dominant arm (Active Comparator): Two ultrasound guided nerve blocks (block of the ulnar and median nerve) on the non-dominant forearm.
  Interventions: Procedure: Non-dominant arm

INTERVENTIONS:
Procedure: Dominant Arm — The volume of local anesthetic used for the block of the ulnar and median nerve will be 5 times the estimated 95% effective dose (ED 95 ) of LA needed to block the nerve relative to the nerve cross-sectional area. The ED 95 for the ulnar nerve has been elucidated to be 0,11ml/mm2. The same ED 95 will be used for the median nerve.
  Arms: Dominant Arm
Procedure: Non-dominant arm — The volume of local anesthetic used for the block of the ulnar and median nerve will be 5 times the estimated 95% effective dose (ED 95 ) of LA needed to block the nerve relative to the nerve cross-sectional area. The ED 95 for the ulnar nerve has been elucidated to be 0,11ml/mm2. The same ED 95 will be used for the median nerve.
  Arms: Non-dominant arm

SUMMARY:
The study aims to describe a correlation between the nerve cross section and the sensory or motor block onset time. Therefore, different nerve cross sections with their Motor and sensory onset times are compared in order to find a correlation.

In the case of discovering a correlation, this could be translated into clinical practice, where a more tailored and individualized approach to performing peripheral nerve blocks would be possible, thus lowering the risks of adverse events occurring.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II, both sexes
* ≥ 18 years old
* < 65 years old
* Written informed consent as documented by signature

Exclusion Criteria:

* Known allergy or hypersensitivity to a study drug or class of drug.
* Severe coagulopathy.
* History of alcohol abuse or the intake of psychotropic drugs.
* Pregnancy.
* Infection at the injection site or a systemic infection.
* Fever of unknown origin.
* Motor or sensory abnormalities in the arm.
* Previous enrollment into the current study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Correlation between nerve cross-section and time to complete sensory block of a nerve | Sensory evaluation will be carried out before the block and every 2 minutes after the start of the injection of LA until complete sensory loss to both cold and pinprick. Expected time frame: 10-60 minutes
  Correlation between the nerve cross-section in mm2 of both nerves (median and ulnar) measured with an ultrasound system and time in minutes from the moment the investigator starts injecting the local anesthetic (LA) around the respective nerves to complete sensory loss in the innervation area of the blocked nerve, assessed by response to light touch, pinprick and cold sensation. This correlation will be expressed in min/ mm2.

SECONDARY OUTCOMES:
Correlation between nerve cross-section and time to complete motor block of a nerve | Motor evaluation will be carried out before the block and every 2 minutes after the start of the injection of LA until complete motor block. Expected time frame: 10-100 minutes
  The correlation between the nerve cross-section area in mm2 of both nerves (median and ulnar) measured with an ultrasound system and time in minutes from the start of the LA injection around the nerve median and ulnar nerves to the respective onset of the motor block, assessed with a numerical scale ranging from 0 to 5 (0-no muscle contraction visible, 5-normal muscle strength, maximal force against resistance and gravity). This correlation will be expressed in min/ mm2.
Correlation between nerve cross-section and the duration of sensory nerve block | The evaluation of the duration of block will start one hour after the determined complete sensory loss and will be tested every 10 minutes until complete resolution of the sensory block. Expected time frame: 10-300 minutes
  The correlation between the nerve cross-section area in mm2 of both nerves (median and ulnar) measured with an ultrasound system and the duration of the respective sensory block in minutes, as reflected by the return of normal sensation in the innervation area of the respective nerve. This correlation will be expressed in min/ mm2.
Correlation between the nerve cross-section and duration of motor nerve block | The evaluation of the duration of sensory block will start one hour after the determined complete motor loss and will be tested every 10 minutes until complete resolution of the motor block. Expected time frame: 10-300min
  The correlation between the nerve cross-section area in mm2 of both nerves (median and ulnar) measured with an ultrasound system and the duration of the respective motor block in minutes, as reflected by the return of normal muscle strength in the innervation area of the respective nerve. This correlation will be expressed in min/ mm2.

CONTACTS AND LOCATIONS:
Overall Officials: José Aguirre, PD Dr Med, Principal Investigator — Der Balgrist
Locations (1):
- Der Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capdevila X, Biboulet P, Morau D, Mannion S, Choquet O. How and why to use ultrasound for regional blockade. Acta Anaesthesiol Belg. 2008;59(3):147-54. PMID 19051446
- [Background] Lewis SR, Price A, Walker KJ, McGrattan K, Smith AF. Ultrasound guidance for upper and lower limb blocks. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD006459. doi: 10.1002/14651858.CD006459.pub3. PMID 26361135
- [Background] Eichenberger U, Stockli S, Marhofer P, Huber G, Willimann P, Kettner SC, Pleiner J, Curatolo M, Kapral S. Minimal local anesthetic volume for peripheral nerve block: a new ultrasound-guided, nerve dimension-based method. Reg Anesth Pain Med. 2009 May-Jun;34(3):242-6. doi: 10.1097/AAP.0b013e31819a7225. PMID 19587623
- [Background] Keplinger M, Marhofer P, Marhofer D, Schroegendorfer K, Haslik W, Zeitlinger M, Mayer CV, Kettner SC. Effective local anaesthetic volumes for sciatic nerve blockade: a clinical evaluation of the ED99. Anaesthesia. 2015 May;70(5):585-90. doi: 10.1111/anae.13013. Epub 2015 Jan 20. PMID 25644578
- [Background] Choi S, McCartney CJ. Evidence Base for the Use of Ultrasound for Upper Extremity Blocks: 2014 Update. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):242-50. doi: 10.1097/AAP.0000000000000155. PMID 25376973
- [Background] Fenten MG, Schoenmakers KP, Heesterbeek PJ, Scheffer GJ, Stienstra R. Effect of local anesthetic concentration, dose and volume on the duration of single-injection ultrasound-guided axillary brachial plexus block with mepivacaine: a randomized controlled trial. BMC Anesthesiol. 2015 Sep 30;15:130. doi: 10.1186/s12871-015-0110-0. PMID 26423050
- [Background] Serradell A, Herrero R, Villanueva JA, Santos JA, Moncho JM, Masdeu J. Comparison of three different volumes of mepivacaine in axillary plexus block using multiple nerve stimulation. Br J Anaesth. 2003 Oct;91(4):519-24. doi: 10.1093/bja/aeg215. PMID 14504153
- [Background] Fredrickson MJ, Abeysekera A, White R. Randomized study of the effect of local anesthetic volume and concentration on the duration of peripheral nerve blockade. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):495-501. doi: 10.1097/AAP.0b013e3182580fd0. PMID 22664978
- [Background] Latzke D, Marhofer P, Zeitlinger M, Machata A, Neumann F, Lackner E, Kettner SC. Minimal local anaesthetic volumes for sciatic nerve block: evaluation of ED 99 in volunteers. Br J Anaesth. 2010 Feb;104(2):239-44. doi: 10.1093/bja/aep368. Epub 2009 Dec 23. PMID 20034967
- [Background] Ecoffey C, Oger E, Marchand-Maillet F, Cimino Y, Rannou JJ, Beloeil H; SOS French Regional Anaesthesia Hotline. Complications associated with 27 031 ultrasound-guided axillary brachial plexus blocks: a web-based survey of 36 French centres. Eur J Anaesthesiol. 2014 Nov;31(11):606-10. doi: 10.1097/EJA.0000000000000063. PMID 24809480
- [Background] Jeng CL, Torrillo TM, Rosenblatt MA. Complications of peripheral nerve blocks. Br J Anaesth. 2010 Dec;105 Suppl 1:i97-107. doi: 10.1093/bja/aeq273. PMID 21148659
- [Background] Hebl JR. The importance and implications of aseptic techniques during regional anesthesia. Reg Anesth Pain Med. 2006 Jul-Aug;31(4):311-23. doi: 10.1016/j.rapm.2006.04.004. No abstract available. PMID 16857551
- [Background] Rotter ML, Hirschl AM, Koller W. Effect of chlorhexidine-containing detergent, non-medicated soap or isopropanol and the influence of neutralizer on bacterial pathogenicity. J Hosp Infect. 1988 Apr;11(3):220-5. doi: 10.1016/0195-6701(88)90100-4. PMID 2899106
- [Background] Marhofer P, Eichenberger U, Stockli S, Huber G, Kapral S, Curatolo M, Kettner S. Ultrasonographic guided axillary plexus blocks with low volumes of local anaesthetics: a crossover volunteer study. Anaesthesia. 2010 Mar;65(3):266-71. doi: 10.1111/j.1365-2044.2010.06247.x. Epub 2010 Jan 29. PMID 20121770